CLINICAL TRIAL: NCT02498535
Title: Prospective, Randomized, Placebo Controlled Trial of the Efficacy and Safety of Inhaled Nitric Oxide (NO) in Cystic Fibrosis (CF) Patients
Brief Title: Efficacy and Safety of Inhaled Nitric Oxide (NO) in Cystic Fibrosis (CF) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for the safety of cystic fibrosis clinical trial subjects due to Covid-19.
Sponsor: Novoteris, LLC (Industry)
Collaborators: Cystic Fibrosis Foundation (Other); Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NO-CF-02E
Record Dates: First submitted 2015-07-12; First posted 2015-07-15 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitric oxide gas at 160 ppm (Experimental): Nitric oxide gas at 160 ppm inhaled four times daily for 30 min delivered with air as the carrier via nasal inhalation for a total of 7.5 days. Total dose of 2400 ppm hours.
  Interventions: Drug: Nitric Oxide 160 ppm
- Breathing 20.3% oxygen (Placebo Comparator): Breathing 20.3% oxygen inhaled four times daily for 30 min delivered with air as the carrier via nasal inhalation for a total of 7.5 days.. 100% nitrogen will be injected into the breathing circuit (instead of 99.5% nitrogen and 0.5% NO).
  Interventions: Drug: Nitric Oxide 160 ppm

INTERVENTIONS:
Drug: Nitric Oxide 160 ppm — Nitric Oxide 160 ppm

SUMMARY:
Prospective, randomized, placebo controlled, phase II clinical study of subjects crossing over from an approved inhaled antibiotic to inhaled nitric oxide as compared to a placebo control arm.

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo controlled, phase II clinical study comparing an investigational drug to a placebo control. Screening data will be reviewed to determine subject eligibility. All subjects including screen failure subjects will be recorded on screening logs at their respective sites. Upon successful completion of all screening procedures, a subject will be considered eligible for enrollment. The subject will be enrolled and randomized in as close a time proximity to the first treatment application as is possible in order to minimize the possibility of dropout while enrolled but before undergoing treatment. With a 1:1 investigational treatment to placebo control, subjects will be randomized to one of the two arms. Subjects in the investigational treatment arm will be administered doses of NO (0.5% NO in 99.5% nitrogen) diluted in room air by inhalation four times daily (30-minute inhalations at least 3 hours apart) for 7.5 days on Days 1, 2, 3, 4, 5, 8, 9, and 10 (three treatments on Days 1 and 10). Subjects in the placebo arm will breathe 100% nitrogen diluted in room air in the same proportion as the investigational arm. Subjects will remain in the clinic for 30 minutes after completing the last treatment of each day. All subjects will be asked to return to the clinic for additional evaluations on Days 15 and 36.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Cystic Fibrosis based on the following criteria:

   * positive sweat chloride 60 mEq/liter (by pilocarpine iontophoresis); and/or
   * a genotype with two identifiable mutations consistent with CF
2. Presence of Pseudomonas aeruginosa, Staphylococcus aureus or Stenotrophomonas maltophilia in the screening sputum culture.
3. Chronic microbial lung colonization (≥6 months) with presence of Pseudomonas aeruginosa, Staphylococcus aureus or Stenotrophomonas maltophilia in at least two (2) sputum cultures in the past year (the screening culture can count as one of the two positive cultures).
4. Ongoing chronic inhaled antibiotic therapy for at least 3 months prior to (screening or baseline).

   • For subjects on cycled therapy, at least 2 cycles of drug need to have been completed prior to baseline.
5. Willing to be off of inhaled antibiotic therapy from Day 1 to Day 15
6. Male or female subjects ≥18 years
7. FEV1 <85% and >35% at screening and baseline
8. SaO2 >90% on room air at screening and baseline
9. Clinically stable with no significant changes in health status within 14 days prior to Baseline
10. Written Informed Consent and HIPAA authorization
11. Non-smoker for at least 6 months prior to screening and agrees not to smoke during the study
12. Chest x-ray within the last six (6) months. If none, a chest x-ray is required before randomization.
13. Willing and able to comply with the treatment schedule and procedures.

Exclusion Criteria:

1. Initiation of any new chronic therapy (e.g., ibuprofen, Pulmozyme®, hypertonic saline, azithromycin, TOBI®, Cayston®) within 4 weeks prior to screening.
2. Use of antibiotics [oral, intravenous (iv), and/or inhaled] for acute respiratory symptoms within 2 weeks prior to baseline.
3. Significant hemoptysis within 30 days prior to screening (≥5 mL of blood in one coughing episode or >30 mL of blood in a 24 hour period)
4. History of colonization with nontuberculosis mycobacterium in sputum culture. The investigator can be guided by the following suggested criteria for a subject to be considered free of colonization:

   * Two respiratory tract cultures negative for NTM in the last year, with no subsequent positive cultures; and
   * these 2 respiratory cultures must be separated by at least 3 months; and
   * one of these two cultures has to have been obtained within the last 6 months
5. Cardiac (left heart) insufficiency (defined as LVEF <35%) at screening
6. Use of a nitric oxide donor agent such as nitroglycerin or drugs known to increase methemoglobin such as lidocaine, prilocaine, benzocaine or dapsone at screening
7. Any of the following abnormal lab values at Screening:

   * Hemoglobin < 10 g/dl
   * Methemoglobn >3%
   * Platelet count <100,000/mm3
   * Prothrombin time international ratio (INR) > 1.5
   * Abnormal liver function defined as any two of the following:
   * ALT >3 x ULN
   * AST >3 x ULN
   * ALP > 3 x ULN
   * GGT > 3 x ULN
   * Abnormal liver function defined as:
   * ALT >5 x ULN
   * AST >5 x ULN
   * Abnormal renal function defined as:
   * Calculated Creatinine Clearance < 50 mL (as calculated by Cockcroft/Gault)
8. For women of child bearing potential:

   * positive pregnancy test at screening or
   * lactating or
   * unwilling to practice a medically acceptable form of contraception from screening to Day 36 (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent)
9. Use of an investigational drug within 30 days prior to screening
10. Intravenous or oral steroids in the 14 days prior to screening
11. Current use of inhaled steroids >500 micrograms twice daily of Fluticasone or equivalent in the 30 days prior to screening
12. Use of supplemental oxygen (daytime or nocturnal) in the 7 days prior to screening
13. Any condition that the Investigator believes would interfere with the intent of this study or would make participation not in the best interest of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 % predicted from baseline to Day 15 | 15 Days
  The primary efficacy variable for this study is absolute change from baseline FEV1% predicted to Day 15. For each subject, the change will be calculated as the FEV1% value minus the baseline FEV1%, i.e., a positive change in FEV1% values will indicate an increase in FEV1% after treatment. The primary endpoint for this trial is the comparison of the mean absolute change from baseline in FEV1% between treatment groups.

SECONDARY OUTCOMES:
Mean absolute change in FEV1% from baseline to Day 15 in the NO group (within group test). | 15 days
  Clinical Measurement of Mean absolute change in FEV1% from baseline to Day 15 in the NO group (within group test).
Mean change in prevalent recovered organisms' sputum CFU g (log 10) from baseline to Days 10, 15 and 36 | 36 days
  Clinical Measurement of Mean change in prevalent recovered organisms' sputum CFU g (log 10) from baseline to Days 10, 15 and 36
Mean change in distance walked in the six-minute walk test from baseline to Days 15 and 36. | 36 days
  Clinical Measurement of Mean change in distance walked in the six-minute walk test from baseline to Days 15 and 36.
Mean absolute change in FEV1 % predicted from baseline to Days 10 and 36. | 36 days
  Clinical Measurement of Mean absolute change in FEV1 % predicted from baseline to Days 10 and 36.
Mean change in FEV1 % predicted (relative) from baseline to Days 10, 15, and 36. | 36 days
  Clinical Measurement of Mean change in FEV1 % predicted (relative) from baseline to Days 10, 15, and 36.
Mean change in FVC from baseline to Days 10, 15 and 36 | 36 days
  Clinical Measurement of Mean change in FVC from baseline to Days 10, 15 and 36
Mean change in FEF25-75 from baseline to Days 10, 15 and 36 | 36 days
  Clinical Measurement of Mean change in FEF25-75 from baseline to Days 10, 15 and 36
Mean change in CFQ-R scores for each domain from baseline to Days 15 and 36 | 36 days
  Clinical Measurement of Mean change in CFQ-R scores for each domain from baseline to Days 15 and 36
Counts of CFRSD-CRISS symptom scores for each symptom from evening prior to Day 1 to each day of the study (Days 1-35) | 35 days
  Clinical Measurement of Counts of CFRSD-CRISS symptom scores for each symptom from evening prior to Day 1 to each day of the study (Days 1-35)
Number of subjects with a relative improvement between baseline and Day 10 in FEV1 % predicted of ≥7.5% | 10 days
  Clinical Measurement of Number of subjects with a relative improvement between baseline and Day 10 in FEV1 % predicted of ≥7.5%
Number of subjects with an absolute improvement in CFQ-R survey scores ≥5 between baseline and Days 15 and 36 | 36 days
  Clinical Measurement of Number of subjects with an absolute improvement in CFQ-R survey scores ≥5 between baseline and Days 15 and 36
Number of subjects with a positive response in the 6 minute walk test at Days 15 and 36 | 36 days
  Clinical Measurement of Number of subjects with a positive response in the 6 minute walk test at Days 15 and 36

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - * Entire USA* The sponsor will provide air transportation and housing to patients that are not located in the area of clinical trial sites. All trial sites can treat adults., Garden Grove, California
  - Children's Hospital of Los Angeles (Adults can be treated here) (Site No. 500), Los Angeles, California
  - Nationwide Children's Hospital (Adults can be treated here) (Site No. 600), Columbus, Ohio
  - Medical University of South Carolina (Site No. 200), Charleston, South Carolina
  - University of Washington Medical Center (Site No. 100), Seattle, Washington
  - Medical College of Wisconsin (Site No. 400), Milwaukee, Wisconsin
- University of British Columbia, St. Paul's Hospital (Site No. 300), Vancouver, B.C., Canada

IPD SHARING:
Plan to Share IPD: No